CLINICAL TRIAL: NCT03257410
Title: A Multi-Center, Prospective, Randomized, Controlled, Open-label, Parallel Study to Evaluate the Safety and Efficacy of the Theranova 400 Dialyzer In End Stage Renal Disease (ESRD) Patients
Brief Title: Theranova 400 Dialyzer In End Stage Renal Disease (ESRD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7905001
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Theranova 400 (Experimental): Three (3) dialysis sessions per week in an in-center setting over 24-week period.
  Interventions: Device: Theranova 400 dialyzer
- Elisio-17H (Active Comparator): Three (3) dialysis sessions per week in an in-center setting over 24-week period.
  Interventions: Device: Elisio-17H dialyzer

INTERVENTIONS:
Device: Theranova 400 dialyzer — Patients should continue with their pre-study hemodialysis prescriptions (in terms of treatment time, blood flow rate and dialysate flow rate) and prescriptions should be kept stable throughout the study.
  Other Names: MCO-Ci 400 Dialyzer; medium cut-off dialysis membrane
  Arms: Theranova 400
Device: Elisio-17H dialyzer — Patients should continue with their pre-study hemodialysis prescriptions (in terms of treatment time, blood flow rate and dialysate flow rate) and prescriptions should be kept stable throughout the study.
  Arms: Elisio-17H

SUMMARY:
The study evaluates the efficacy and safety of the Theranova 400 dialyzer compared with Elisio-17 H dialyzer in end stage renal disease patients receiving hemodialysis treatment. Efficacy will be determined by the removal of middle molecules (with different molecular size) from the blood compartment. Safety will be evaluated by maintaining pre-dialysis serum albumin levels and other safety events including laboratory tests and adverse events.

Patients will undergo 3 dialysis sessions per week, for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients age 22 and older, or between ages 18 and 21 with a weight ≥ 40kg.
* Clinically stable as judged by the treating physician and as demonstrated by stable medical history for 30 days prior to enrollment, physical examination, and laboratory testing.
* Hemodialysis therapy with high-flux dialyzers for at least 3 months immediately prior to study enrollment and expected to survive for the next 12 months.
* Expected to maintain an acceptable urea clearance (Kt/V) with a dialyzer of an approximate surface area of 1.7 m2.
* Currently being dialyzed at an in-center setting, on a schedule of 3 times per week.
* Able to give informed consent after an explanation of the proposed study, and who are willing to comply with the study requirements for therapy during the entire study treatment period.
* Have a stable functioning vascular access (arteriovenous fistula, graft, or dual lumen tunneled catheter); stable access will be confirmed by observed Kt/V >= 1.2 for past 2 measurements, and/or achievement of within 15% the prescribed blood flow rate over 3 treatments prior to study entry.

Exclusion Criteria:

* Are female and pregnant, lactating, or planning to become pregnant during the study period. Note: Female subjects of childbearing potential, defined as a woman <55 years old who has not had a partial or full hysterectomy or oophorectomy, must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at screening. Subjects of childbearing potential must use a medically acceptable means of contraception during their participation in the study.
* Have chronic liver disease.
* Have a known paraprotein-associated disease.
* Have known bleeding disorders (e.g., gastrointestinal bleed, colonic polyps, small bowel angiodysplasia, and active peptic ulcers).
* Have had a major bleeding episode (i.e. soft tissue bleeding, blood in stool, prolonged nose bleeds, joint damage, retinal bleeding, extensive mucosal bleeding, exsanguination, cerebral hemorrhage) ≤ 12 weeks prior to randomization.
* Have had a blood (red blood cell) transfusion ≤ 12 weeks prior to randomization.
* Have had an acute infection ≤ 4 weeks prior to randomization.
* Have active cancer, except for basal cell or squamous cell skin cancer.
* Have a known serum κ/λ FLC ratio that is less than 0.37, or greater than 3.1.b
* Have a known monoclonal gammopathy (monoclonal gammopathy of uncertain significance, smoldering [asymptomatic] multiple myeloma, symptomatic multiple myeloma, plasmacytomas, or plasma cell leukemia).
* Have a known polyclonal gammopathy (connective tissue disease, liver disease, chronic infection, lymphoproliferative disorder, or other hematologic condition).
* Have a positive serology test for human immunodeficiency virus or hepatitis infection.
* Have a significant psychiatric disorder or mental disability.
* Are scheduled for planned interventions requiring hospitalization > 1 week.
* Are scheduled for living-donor transplantation within the study period + 3 months, plan to change to PD therapy within the next 9 months, plan to change to a home hemodialysis treatment, or plan to relocate to an area where no study center is located.
* Are currently participating in another interventional clinical study or has participated in another interventional clinical study in the past 3 months.
* Have a history of non-compliance with HD as assessed by an investigator.
* Have had a major cardiovascular or cerebrovascular event within 3 months of study entry.
* Have a history with consistent evidence of intradialytic hypotension.
* Have uncontrolled (systolic BP > 180 mmHg) hypertension.
* Have had adverse reactions to dialyzer materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - DaVita Corona, Corona, California
  - DaVita Riverside, Riverside, California
  - DaVita Inc, Greater Hartford Nephrology, Bloomfield, Connecticut
  - DaVita Inc., Waterbury Dialysis, Middlebury, Connecticut
  - Dialysis Center, Inc. Albany, Albany, Georgia
  - Dialysis Center, Inc. Boston, Boston, Massachusetts
  - Dialysis Center, Inc. Kidney Associates of Kansas City, Belton, Missouri
  - Dialysis Center of Lincoln, Lincoln, Nebraska
  - DaVita Five Star Dialysis Center, Las Vegas, Nevada
  - DaVita Inc., South Las Vegas Dialysis, Las Vegas, Nevada
  - Dialysis Center, Inc. North Brunswick, North Brunswick, New Jersey
  - DaVita Inc., Bronx Dialysis Center, The Bronx, New York
  - Dialysis Center, Inc. Philidelphia, Philadelphia, Pennsylvania
  - Dialysis Center, Inc. Holston River Clinic, Knoxville, Tennessee
  - DaVita Inc., Transmountain Dialysis, El Paso, Texas
  - DaVita Inc., Medical Center Dialysis, Houston, Texas
  - DaVita Renal Center of Lewisville, Lewisville, Texas
  - DaVita Inc., Northwest Medical Center Dialysis, San Antonio, Texas
  - DaVita Floyd Curl Dialysis, San Antonio, Texas
  - DaVita Inc., Norfolk Dialysis, Chesapeake, Virginia

REFERENCES:
- [Result] Weiner DE, Falzon L, Skoufos L, Bernardo A, Beck W, Xiao M, Tran H. Efficacy and Safety of Expanded Hemodialysis with the Theranova 400 Dialyzer: A Randomized Controlled Trial. Clin J Am Soc Nephrol. 2020 Sep 7;15(9):1310-1319. doi: 10.2215/CJN.01210120. Epub 2020 Aug 25. PMID 32843372
- See also: Related Info — https://cjasn.asnjournals.org/content/15/9/1310

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theranova 400 | Elisio-17H
Started | 86 | 86
Completed | 65 | 65
Not Completed | 21 | 21
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Renal transplantation | 2 | 0
Not completed — Switch to peritoneal dialysis | 1 | 0
Not completed — Death | 3 | 2
Not completed — Change to another dialysis center | 2 | 2
Not completed — Missing 3 consecutive study treatments | 5 | 6
Not completed — Miscellaneous | 2 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theranova 400 | Elisio-17H | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (13.52) | 59.7 (12.4) | 59.1 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 67
  Male | 54 | 51 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Black or African American | 33 | 35 | 68
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  White | 40 | 42 | 82
  Other | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 86 | 172

OUTCOME MEASURES:

1. Primary Outcome: Reduction Ratio of Lambda Immunoglobulin FLC at Week 24
Description: FLC=free light chains
Time Frame: Week 24
Population: Full Analysis Set. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 82 | 79
percentage ratio | 32.156 (12.602) | 17.514 (12.7235)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; If the lower bound of the two-sided 95% confidence interval around the difference between Theranova 400 and Elisio-17H is > 0 then superiority will be demonstrated; Test type: Superiority; Mean Difference (Final Values) = 14.828, 95% CI 2-sided [10.501 to 19.156] — Method=ANCOVA

2. Primary Outcome: Pre-dialysis Serum Level of Albumin at Week 24
Time Frame: Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 84 | 83
g/dL | 4.030 (0.2843) | 4.018 (0.3935)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Non-Inferiority — If the lower bound of the two-sided 95% confidence interval around the mean estimated treatment difference between Theranova 400 and Elisio 17H is > -0.1765 g/dL then non-inferiority can be claimed. If the lower bound of the two-sided 95% confidence interval is > 0, then superiority may be concluded; ANCOVA; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.098 to 0.069]

3. Secondary Outcome: Reduction Ratio of Lambda Immunoglobulin FLC at Week 4 and Week 24
Description: FLC=free light chains
Time Frame: Week 4 and Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 80 | 75
  Week 4 | 39.3 (14.487) | 19.88 (11.394)
  Week 24: number analyzed (Participants) | 63 | 65
  Week 24 | 33.29 (10.96) | 17.19 (12.863)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p < 0.0001, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = 19.42, Standard Error of Mean 2.103
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p < 0.0001, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = 16.10, Standard Error of Mean 2.115

4. Secondary Outcome: Reduction Ratio of Complement Factor D
Description: CFD=complement factor D
Time Frame: Week 4 and 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 83 | 76
  Week 4 | 36.78 (26.499) | 11.71 (27.71)
  Week 24: number analyzed (Participants) | 62 | 65
  Week 24 | 38.09 (11.233) | 14.55 (11.298)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p < 0.0001, MMRM; Mean Difference (Final Values) = 25.07, Standard Error of Mean 4.300
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p < 0.0001, MMRM; Mean Difference (Final Values) = 23.54, Standard Error of Mean 2.000

5. Secondary Outcome: Reduction Ratio of κ FLC
Description: κ FLC = Kappa Free light chains
Time Frame: Week 4 and 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 80 | 75
  Week 4 | 65.63 (18.566) | 49.74 (15.111)
  Week 24: number analyzed (Participants) | 63 | 65
  Week 24 | 59.27 (13.068) | 43.91 (14.882)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p < 0.0001, MMRM; Mean Difference (Final Values) = 15.89, Standard Error of Mean 2.730
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p < 0.0001, MMRM; Mean Difference (Final Values) = 15.36, Standard Error of Mean 2.479

6. Secondary Outcome: Reduction Ratio of Interleukin 6
Description: IL-6=interleukin 6
Time Frame: Week 4 and 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 80 | 78
  Week 4 | -4.62 (49.378) | -22.21 (69.618)
  Week 24: number analyzed (Participants) | 63 | 65
  Week 24 | -0.85 (46.214) | -14.83 (43.574)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p = 0.0684, MMRM; Mean Difference (Final Values) = 17.59, Standard Error of Mean 9.583
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.0806, MMRM; Mean Difference (Final Values) = 13.98, Standard Error of Mean 7.937

7. Secondary Outcome: Reduction Ratio of Tumor Necrosis Factor Alpha
Description: TNFα=tumor necrosis factor alpha
Time Frame: Week 4 and 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 80 | 78
  Week 4 | 47.29 (9.966) | 37.9 (8.892)
  Week 24: number analyzed (Participants) | 63 | 65
  Week 24 | 44.48 (10.215) | 34.52 (10.673)

8. Secondary Outcome: Reduction Ratio of β2-microglobulin
Description: β2=beta 2
Time Frame: Week 4 and 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage ratio
  Week 4: number analyzed (Participants) | 78 | 76
  Week 4 | 75.67 (8.2) | 64.86 (8.903)
  Week 24: number analyzed (Participants) | 63 | 65
  Week 24 | 73.64 (10.426) | 65.41 (9.428)

9. Secondary Outcome: Change From Baseline in Pre-dialysis β2-microglobulin at Week 24
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 64
mg/L | -3.95 (5.614) | -1.16 (6.128)

10. Secondary Outcome: Kt/Vurea
Description: Kt/Vurea = Dimensionless number used to quantify hemodialysis and peritoneal dialysis adequacy.
Time Frame: Week 4, 8, 12, 16, 20, 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: Kt/Vurea
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
Kt/Vurea
  Week 4: number analyzed (Participants) | 78 | 76
  Week 4 | 1.58 (0.266) | 1.58 (0.427)
  Week 8: number analyzed (Participants) | 76 | 76
  Week 8 | 1.62 (0.288) | 1.51 (0.316)
  Week 12: number analyzed (Participants) | 77 | 70
  Week 12 | 1.58 (0.294) | 1.55 (0.328)
  Week 16: number analyzed (Participants) | 69 | 70
  Week 16 | 1.56 (0.268) | 1.59 (0.48)
  Week 20: number analyzed (Participants) | 66 | 69
  Week 20 | 1.57 (0.297) | 1.55 (0.371)
  Week 24: number analyzed (Participants) | 62 | 65
  Week 24 | 1.51 (0.31) | 1.54 (0.467)

11. Secondary Outcome: Change From Baseline in Pre-dialysis Serum Albumin by Visit
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
g/dL
  Week 4: number analyzed (Participants) | 80 | 77
  Week 4 | -0.08 (0.244) | 0 (0.203)
  Week 8: number analyzed (Participants) | 78 | 77
  Week 8 | -0.11 (0.254) | 0.00 (0.216)
  Week 12: number analyzed (Participants) | 77 | 72
  Week 12 | -0.12 (0.289) | -0.04 (0.229)
  Week 16: number analyzed (Participants) | 72 | 71
  Week 16 | -0.13 (0.335) | -0.03 (0.315)
  Week 20: number analyzed (Participants) | 66 | 69
  Week 20 | -0.08 (0.279) | 0.02 (0.258)
  Week 24: number analyzed (Participants) | 64 | 65
  Week 24 | 0.01 (0.250) | 0.04 (0.256)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p = 0.0347, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.07, Standard Error of Mean 0.033
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 8; Test type: Other; p = 0.0036, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.10, Standard Error of Mean 0.033
Statistical Analysis 3: Comparison: Theranova 400 vs Elisio-17H; Week 12; Test type: Other; p = 0.129, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.040
Statistical Analysis 4: Comparison: Theranova 400 vs Elisio-17H; Week 16; Test type: Other; p = 0.1149, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.08, Standard Error of Mean 0.052
Statistical Analysis 5: Comparison: Theranova 400 vs Elisio-17H; Week 20; Test type: Other; p = 0.0688, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.08, Standard Error of Mean 0.044
Statistical Analysis 6: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.6097, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.02, Standard Error of Mean 0.042

12. Secondary Outcome: Change From Baseline in Pre-dialysis Factor VII by Visit
Time Frame: Baseline, Week 12, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage activity
  Week 12: number analyzed (Participants) | 73 | 70
  Week 12 | 3.59 (24.057) | 7.79 (27.798)
  Week 24: number analyzed (Participants) | 60 | 63
  Week 24 | 0.38 (34.572) | 9.19 (48.575)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 12; Test type: Other; p = 0.1472, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -6.32, Standard Error of Mean 4.336
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.1207, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -11.18, Standard Error of Mean 7.154

13. Secondary Outcome: Change From Baseline in Pre-dialysis Protein C by Visit
Time Frame: Baseline, Week 12, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percentage activity
  Week 12: number analyzed (Participants) | 75 | 70
  Week 12 | 1.12 (15.711) | 1.76 (16.378)
  Week 24: number analyzed (Participants) | 63 | 63
  Week 24 | 0.14 (19.376) | -1.78 (18.781)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 12; Test type: Other; p = 0.9775, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.07, Standard Error of Mean 2.488
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.5538, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = 1.72, Standard Error of Mean 2.905

14. Secondary Outcome: Change From Baseline in Pre-dialysis Vitamin A by Visit
Time Frame: Baseline, Week 4, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
μmol/L
  Week 4: number analyzed (Participants) | 75 | 74
  Week 4 | -0.29 (0.983) | -0.04 (0.939)
  Week 24: number analyzed (Participants) | 59 | 61
  Week 24 | -0.33 (0.832) | -0.15 (1.096)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p = 0.1100, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.23, Standard Error of Mean 0.146
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.4607, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.11, Standard Error of Mean 0.153

15. Secondary Outcome: nPNA (nPCR)
Description: nPNA=normalized Protein equivalent of Nitrogen Appearance, and nPCR=normalized Protein Catabolic Rate.
Time Frame: Week 4, 8, 12, 16, 20, 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/kg/d
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
g/kg/d
  Week 4: number analyzed (Participants) | 78 | 76
  Week 4 | 0.983 (0.2473) | 1.056 (0.3088)
  Week 8: number analyzed (Participants) | 75 | 75
  Week 8 | 1.013 (0.2380) | 1.023 (0.2936)
  Week 12: number analyzed (Participants) | 77 | 70
  Week 12 | 0.971 (0.2573) | 1.030 (0.2664)
  Week 16: number analyzed (Participants) | 69 | 70
  Week 16 | 1.022 (0.2869) | 0.971 (0.2881)
  Week 20: number analyzed (Participants) | 66 | 69
  Week 20 | 0.988 (0.2666) | 1.024 (0.3366)
  Week 24: number analyzed (Participants) | 62 | 65
  Week 24 | 0.947 (0.2450) | 1.012 (0.2891)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 4; Test type: Other; p = 0.0791, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.0787, Standard Error of Mean 0.04454
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 8; Test type: Other; p = 0.9505, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.0027, Standard Error of Mean 0.04302
Statistical Analysis 3: Comparison: Theranova 400 vs Elisio-17H; Week 12; Test type: Other; p = 0.1521, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.0615, Standard Error of Mean 0.04271
Statistical Analysis 4: Comparison: Theranova 400 vs Elisio-17H; Week 16; Test type: Other; p = 0.2489, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = 0.0538, Standard Error of Mean 0.04652
Statistical Analysis 5: Comparison: Theranova 400 vs Elisio-17H; Week 20; Test type: Other; p = 0.4936, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.0345, Standard Error of Mean 0.05025
Statistical Analysis 6: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.1497, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.0663, Standard Error of Mean 0.04580

16. Secondary Outcome: Change From Baseline in Pre-dialysis Factor II by Visit
Description: Factor II (Prothrombin)
Time Frame: Baseline, Week 12, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percent activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
percent activity
  Week 12: number analyzed (Participants) | 73 | 70
  Week 12 | 3.45 (11.507) | 3.19 (13.284)
  Week 24: number analyzed (Participants) | 60 | 63
  Week 24 | 3.85 (11.678) | 5.78 (15.394)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Week 12; Test type: Other; p = 0.9001, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -0.25, Standard Error of Mean 2.012
Statistical Analysis 2: Comparison: Theranova 400 vs Elisio-17H; Week 24; Test type: Other; p = 0.3279, Mixed-effect Model Repeated Measurement; Mean Difference (Final Values) = -2.33, Standard Error of Mean 2.372

17. Secondary Outcome: Change From Baseline in Sodium (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline and Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.20 (3.192) | 0.00 (3.671)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.6576, ANCOVA; Mean Difference (Final Values) = 0.20, Standard Error of Mean 0.452

18. Secondary Outcome: Change From Baseline in Potassium (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline and Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | 0.08 (0.727) | -0.23 (0.665)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0058, ANCOVA; Mean Difference (Final Values) = 0.29, Standard Error of Mean 0.104

19. Secondary Outcome: Change From Baseline in Calcium (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.06 (0.154) | -0.02 (0.151)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.034, ANCOVA; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.023

20. Secondary Outcome: Change From Baseline in Phosphate (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.03 (0.438) | -0.19 (0.500)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0285, ANCOVA; Mean Difference (Final Values) = 0.16, Standard Error of Mean 0.071

21. Secondary Outcome: Change From Baseline in Chloride (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | 0.09 (3.488) | 0.43 (4.108)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.9069, ANCOVA; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.513

22. Secondary Outcome: Change From Baseline in Bicarbonate (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 73
mmol/L | 1.31 (3.053) | 1.37 (3.080)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.8413, ANCOVA; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.443

23. Secondary Outcome: Change From Baseline in Glucose (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
mmol/L | -0.20 (2.197) | 0.47 (2.858)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0125, ANCOVA; Mean Difference (Final Values) = -0.97, Standard Error of Mean 0.382

24. Secondary Outcome: Change From Baseline in Prothrombin Time (Sec) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: Sec
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 72 | 73
Sec | -0.04 (4.016) | -0.49 (6.305)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.6891, ANCOVA; Mean Difference (Final Values) = 0.22, Standard Error of Mean 0.561

25. Secondary Outcome: Change From Baseline in Prothrombin Intl. Normalized Ratio at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 73 | 76
ratio | -0.01 (0.341) | -0.05 (0.527)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.6043, ANCOVA; Mean Difference (Final Values) = 0.02, Standard Error of Mean 0.047

26. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (Sec) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: Sec
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 69 | 72
Sec | -0.82 (16.682) | -0.96 (15.424)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5067, ANCOVA; Mean Difference (Final Values) = 1.39, Standard Error of Mean 2.080

27. Secondary Outcome: Change From Baseline in Hematocrit (L/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 60 | 54
L/L | 0.03 (0.055) | 0.01 (0.042)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0297, ANCOVA; Mean Difference (Net) = 0.02, Standard Error of Mean 0.009

28. Secondary Outcome: Change From Baseline in Hemoglobin (g/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 73 | 72
g/L | 2.74 (15.569) | -0.11 (11.221)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1325, ANCOVA; Mean Difference (Final Values) = 3.24, Standard Error of Mean 2.140

29. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin (pg) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 73 | 72
pg | -0.12 (1.079) | -0.35 (1.153)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2304, ANCOVA; Mean Difference (Final Values) = 0.22, Standard Error of Mean 0.186

30. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular HGB Concentration (g/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 71 | 65
g/L | -18.54 (16.053) | -15.12 (21.075)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5785, ANCOVA; Mean Difference (Final Values) = -1.59, Standard Error of Mean 2.846

31. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume (fL) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 60 | 54
fL | 4.88 (5.371) | 1.93 (4.778)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0067, ANCOVA; Mean Difference (Final Values) = 2.55, Standard Error of Mean 0.918

32. Secondary Outcome: Change From Baseline in Platelets at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 72 | 73
10^9 cells/L | -8.65 (41.711) | 7.99 (49.215)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0434, ANCOVA; Mean Difference (Final Values) = -14.93, Standard Error of Mean 7.314

33. Secondary Outcome: Change From Baseline in Erythrocytes at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 73 | 73
10^12 cells/L | 0.10 (0.482) | 0.04 (0.365)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.3281, ANCOVA; Mean Difference (Final Values) = 0.07, Standard Error of Mean 0.070

34. Secondary Outcome: Change From Baseline in Leukocytes at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 73 | 72
10^9 cells/L | -0.22 (1.640) | 0.49 (2.464)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0463, ANCOVA; Mean Difference (Final Values) = -0.67, Standard Error of Mean 0.334

35. Secondary Outcome: Change From Baseline in Basophils (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: % of total white blood count (WBC)
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
% of total white blood count (WBC) | 0.05 (0.369) | -0.02 (0.408)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1925, ANCOVA; Mean Difference (Final Values) = 0.08, Standard Error of Mean 0.060

36. Secondary Outcome: Change From Baseline in Eosinophils (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: % of total WBC
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
% of total WBC | 0.17 (3.259) | -0.29 (2.397)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2569, ANCOVA; Mean Difference (Final Values) = 0.44, Standard Error of Mean 0.389

37. Secondary Outcome: Change From Baseline in Lymphocytes (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: % of total WBC
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
% of total WBC | 0.14 (6.979) | -0.69 (8.052)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5709, ANCOVA; Mean Difference (Final Values) = 0.63, Standard Error of Mean 1.104

38. Secondary Outcome: Change From Baseline in Monocytes (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: % of total WBC
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
% of total WBC | -0.49 (2.261) | -1.07 (3.479)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.217, ANCOVA; Mean Difference (Final Values) = 0.51, Standard Error of Mean 0.412

39. Secondary Outcome: Change From Baseline in Neutrophils (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: % of total WBC
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 76 | 75
% of total WBC | 0.16 (8.744) | 1.98 (9.485)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2386, ANCOVA; Mean Difference (Final Values) = -1.53, Standard Error of Mean 1.292

40. Secondary Outcome: Change From Baseline in Pre-Dialysis Blood Urea Nitrogen (mmol Urea/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol urea/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 63 | 64
mmol urea/L | -1.82 (5.299) | -0.69 (4.784)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1769, ANCOVA; Mean Difference (Final Values) = -1.14, Standard Error of Mean 0.840

41. Secondary Outcome: Change From Baseline in Post-Dialysis Blood Urea Nitrogen (mmol Urea/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol urea/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 61 | 65
mmol urea/L | -0.53 (2.360) | -0.57 (2.066)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.8102, ANCOVA; Mean Difference (Final Values) = -0.09, Standard Error of Mean 0.360

42. Secondary Outcome: Change From Baseline in BUN Reduction Ratio at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: no unit
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 60 | 63
no unit | 0.33 (9.298) | 0.68 (8.963)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.9672, ANCOVA; Mean Difference (Final Values) = -0.06, Standard Error of Mean 1.501

43. Secondary Outcome: Change From Baseline in Creatinine (μmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
μmol/L | -17.45 (160.343) | -36.44 (153.168)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2697, ANCOVA; Mean Difference (Final Values) = 27.34, Standard Error of Mean 24.623

44. Secondary Outcome: Kt/Vurea by Visit
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: no unit
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 86 | 86
no unit
  Week 4: number analyzed (Participants) | 78 | 76
  Week 4 | 1.58 (0.266) | 1.58 (0.427)
  Week 8: number analyzed (Participants) | 76 | 76
  Week 8 | 1.62 (0.288) | 1.51 (0.316)
  Week 12: number analyzed (Participants) | 77 | 70
  Week 12 | 1.58 (0.294) | 1.55 (0.328)
  Week 16: number analyzed (Participants) | 69 | 70
  Week 16 | 1.56 (0.268) | 1.59 (0.480)
  Week 20: number analyzed (Participants) | 66 | 69
  Week 20 | 1.57 (0.297) | 1.55 (0.371)
  Week 24: number analyzed (Participants) | 62 | 65
  Week 24 | 1.51 (0.310) | 1.54 (0.467)

45. Secondary Outcome: Change From Baseline in Vitamin A (μmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 58 | 58
μmol/L | -0.35 (0.826) | -0.01 (0.899)

46. Secondary Outcome: Change From Baseline in Cholesterol (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.19 (0.766) | -0.24 (0.705)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.7189, ANCOVA; Mean Difference (Final Values) = 0.04, Standard Error of Mean 0.115

47. Secondary Outcome: Change From Baseline in HDL Cholesterol (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | 0.04 (0.266) | -0.03 (0.276)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.097, ANCOVA; Mean Difference (Final Values) = 0.07, Standard Error of Mean 0.044

48. Secondary Outcome: Change From Baseline in LDL Cholesterol (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.07 (0.663) | -0.18 (0.807)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.4513, ANCOVA; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.113

49. Secondary Outcome: Change From Baseline in Triglycerides (mmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
mmol/L | -0.15 (0.661) | -0.02 (0.672)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0733, ANCOVA; Mean Difference (Final Values) = -0.18, Standard Error of Mean 0.100

50. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (U/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 74 | 73
U/L | -1.97 (37.783) | 2.19 (32.725)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5326, ANCOVA; Mean Difference (Final Values) = -3.42, Standard Error of Mean 5.467

51. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (U/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 70 | 70
U/L | -2.17 (8.168) | -0.51 (8.018)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.3042, ANCOVA; Mean Difference (Final Values) = -1.11, Standard Error of Mean 1.076

52. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (U/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 69 | 69
U/L | -0.75 (6.816) | -0.01 (5.870)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5534, ANCOVA; Mean Difference (Final Values) = -0.58, Standard Error of Mean 0.976

53. Secondary Outcome: Change From Baseline in Direct Bilirubin (μmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 3 | 7
μmol/L | 1.53 (2.603) | 0.23 (1.107)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2958, ANCOVA; Mean Difference (Final Values) = 1.34, Standard Error of Mean 1.181

54. Secondary Outcome: Change From Baseline in Bilirubin (μmol/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 72 | 73
μmol/L | -1.06 (2.960) | -0.66 (2.040)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0998, ANCOVA; Mean Difference (Final Values) = -0.63, Standard Error of Mean 0.377

55. Secondary Outcome: Change From Baseline in Gamma Glutamyl Transferase (U/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 74 | 73
U/L | -0.66 (22.587) | -1.68 (21.724)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.9952, ANCOVA; Mean Difference (Final Values) = 0.02, Standard Error of Mean 3.176

56. Secondary Outcome: Change From Baseline in Protein (g/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 74 | 73
g/L | -1.55 (4.576) | -0.95 (4.223)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.3063, ANCOVA; Mean Difference (Final Values) = -0.71, Standard Error of Mean 0.693

57. Secondary Outcome: Change From Baseline in Globulin (g/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 74 | 73
g/L | -2.07 (3.635) | -1.27 (3.216)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1098, ANCOVA; Mean Difference (Final Values) = -0.85, Standard Error of Mean 0.529

58. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (mg/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 47 | 49
mg/L | -0.96 (4.168) | -0.40 (4.600)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0766, ANCOVA; Mean Difference (Final Values) = -1.44, Standard Error of Mean 0.797

59. Secondary Outcome: Change From Baseline in Prothrombin Activity (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 68 | 67
percentage activity | 3.85 (11.678) | 5.78 (15.394)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.2886, ANCOVA; Mean Difference (Final Values) = -2.58, Standard Error of Mean 2.410

60. Secondary Outcome: Change From Baseline in Albumin (g/dL) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 75 | 74
g/dL | 0.01 (0.250) | 0.04 (0.256)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.4513, ANCOVA; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.042

61. Secondary Outcome: Change From Baseline in Factor XIV Activity (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 71 | 67
percentage activity | 0.14 (19.376) | -1.78 (18.781)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.5992, ANCOVA; Mean Difference (Final Values) = 1.56, Standard Error of Mean 2.960

62. Secondary Outcome: Change From Baseline in Tumor Necrosis Factor (pg/mL) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 65
pg/mL | -0.47 (1.999) | 0.08 (1.645)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.3836, ANCOVA; Mean Difference (Final Values) = -0.26, Standard Error of Mean 0.290

63. Secondary Outcome: Change From Baseline in Factor VII Activity (%) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: percentage activity
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 67 | 67
percentage activity | 0.38 (34.572) | 9.19 (48.575)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0769, ANCOVA; Mean Difference (Final Values) = -13.07, Standard Error of Mean 7.284

64. Secondary Outcome: Change From Baseline in Lambda Light Chain, Free (mg/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 65
mg/L | -19.40 (31.635) | 1.75 (29.946)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -19.56, Standard Error of Mean 5.170

65. Secondary Outcome: Change From Baseline in Interleukin 6 (pg/mL) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 65
pg/mL | 0.20 (5.449) | 1.64 (6.473)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1825, ANCOVA; Mean Difference (Final Values) = -1.39, Standard Error of Mean 1.039

66. Secondary Outcome: Change From Baseline in Complement Factor D (mcg/mL) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 62 | 65
mcg/mL | 0.13 (4.742) | 1.89 (4.838)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0957, ANCOVA; Mean Difference (Final Values) = -1.24, Standard Error of Mean 0.737

67. Secondary Outcome: Change From Baseline in Kappa Light Chain, Free (mg/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 65
mg/L | -84.81 (97.359) | -43.01 (75.677)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.0012, ANCOVA; Mean Difference (Final Values) = -34.02, Standard Error of Mean 10.230

68. Secondary Outcome: Change From Baseline in Beta-2 Microglobulin (mg/L) at End of Study (up to Week 24)
Time Frame: Baseline, Week 24
Population: FAS. Number of subjects (n) with evaluable data is shown.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Theranova 400 | Elisio-17H
Number analyzed (Participants) | 64 | 64
mg/L | -3.95 (5.614) | -1.16 (6.128)
Statistical Analysis 1: Comparison: Theranova 400 vs Elisio-17H; Test type: Other; p = 0.1824, ANCOVA; Mean Difference (Final Values) = -1.17, Standard Error of Mean 0.859

ADVERSE EVENTS:
Time Frame: AEs/SAEs were collected after the informed consent was signed and throughout the study (week 24), until the end of study visit (week 25-26).
Arm/Group | Theranova 400 | Elisio-17H
All-Cause Mortality (participants affected / at risk) | 3/86 | 3/85
Serious Adverse Events (participants affected / at risk) | 15/86 | 23/85
Other Adverse Events (participants affected / at risk) | 14/86 | 11/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theranova 400 (N=86) | Elisio-17H (N=85)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (2)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (2)
PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
GRAFT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CALCIPHYLAXIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ANAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theranova 400 (N=86) | Elisio-17H (N=85)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 3 (3) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right of prior review and approval of data from this study relative to the potential release of proprietary information to any publication or for any presentation.

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03257410/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03257410/SAP_001.pdf